CLINICAL TRIAL: NCT04916691
Title: Erector Spinae Plane Block for Rib Fractures: A Pilot Study
Brief Title: Ultrasound-guided Erector Spinae Plane Blocks
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel Stephens, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-007896
Record Dates: First submitted 2021-05-20; First posted 2021-06-07 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPSB for rib fractures (Other): EPSB for rib fractures
  Interventions: Procedure: EPSB for rib fractures; Drug: Ropivacaine

INTERVENTIONS:
Procedure: EPSB for rib fractures — EPSB for rib fractures
Drug: Ropivacaine — Standard of care weight-based optimal Ropivacaine dosing for ESPB

SUMMARY:
The purpose of this study is to determine the feasibility of using the ultrasound-guided erector spinae plane blocks to provide additional pain relief to patients with rib fractures in the Emergency Department (ED) and Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older.
* Patients with one or more acute traumatic rib fractures.

Exclusion Criteria:

* Inability to position appropriately.
* Unconscious or heavily sedated.
* Patients who are critically ill such that care should not be delayed for regional anesthesia.
* Patients under the age of 18 years old.
* Vulnerable populations including prison inmates and pregnant patients.
* Overlying skin infection, wound, or dressing/equipment (i.e., Chest tube).
* Inability to visualize target anatomy or by ultrasound or anatomy prohibitive for other reasons to perform procedure successfully.
* Known or documented allergy to ropivacaine or other amide local anesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Procedural success rate | 12 months
  Measuring the Number of successful ESPB procedures performed in the ED and ICU

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stephens, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials